CLINICAL TRIAL: NCT02640534
Title: Investigation of Metformin in Patients With Castration Resistant Prostate Cancer in Combination With Enzalutamide vs. Enzalutamide Alone (IMPROVE TRIAL): A Randomized, Open Label, Phase II Trial
Brief Title: Investigation of Metformin in Patients With Castration Resistant Prostate Cancer in Combination With Enzalutamide vs. Enzalutamide Alone
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision is based on the fact that with the current follow up of around 10 years, the relevant secondary endpoints can adequately be addressed according to protocol. The addition of follow up data will not significantly impact these results.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 08/14 - IMPROVE
Record Dates: First submitted 2015-12-22; First posted 2015-12-29 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Cancer of the Prostate; Prostate Cancer
Keywords: Prostate cancer; Cancer of the prostate; Metformin; Enzalutamide; Xtandi; castration resistant prostate cancer; phase II; Androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enzalutamide + Metformin (Experimental): Enzalutamide 160 mg od + metformin 850 mg bid until disease progression
  Interventions: Drug: Enzalutamide; Drug: Metformin
- Enzalutamide (Active Comparator): Enzalutamide 160 mg od until disease progression
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide 160 mg od until disease progression
Drug: Metformin — 850 mg bid until disease progression
  Arms: Enzalutamide + Metformin

SUMMARY:
The purpose of this trial is to test if the combination of enzalutamide and metformin in patients with castration resistant prostate cancer CRPC progressing on androgen deprivation therapy ADT is more effective compared to enzalutamide alone. The half of the patients will receive the experimental treatment combination, enzalutamide and metformin, while the other half will receive enzalutamide alone.

DETAILED DESCRIPTION:
One in seven men will be diagnosed with cancer of the prostate during his lifetime . Accordingly, prostate cancer (PC) is the most common cancer amongst men in the western world and worldwide. PC ranks second in cancer incidence and sixth in cancer mortality in men. The current standard of care for patients with metastatic castration resistant prostate cancer (mCRPC) and disease progression is either treatment with abiraterone acetate and prednisone in asymptomatic or mildly symptomatic patients without visceral metastases, or treatment with docetaxel in more symptomatic patients and in the presence of visceral metastases.

Rothemundt et al. previously demonstrated favorable effects of metformin in a phase II trial: it yields objective Prostate specific antigen PSA responses and may induce disease stabilization and improve metabolic endpoints in patients with CRPC. Therefore addition of metformin to enzalutamide might have positive impact on tumor progression, on body composition, and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration and prior to any trial-related investigations
* Histologically or cytological confirmed adenocarcinoma of the prostate without small cell carcinoma or small cell components
* Asymptomatic or minimally symptomatic patients in relation to disease
* Metastatic adenocarcinoma of the prostate documented by imaging (CT/MRI and/or bone scan)
* Ongoing androgen deprivation therapy with Gonadotropin-releasing hormone GnRH analogues or bilateral orchiectomy (i.e. surgical or medical castration)
* Total testosterone levels ≤ 1.7 nmol/L (corresponding to ≤ 50 ng/dL)
* Tumor progression at the time of registration, defined as per protocol.
* Completed baseline QoL and pain questionnaires
* Male patients ≥ 18 years
* WHO performance status 0-2
* Adequate hematologic values: hemoglobin ≥ 90 g/L, neutrophils ≥ 1.0 x 109/L, platelets ≥ 75 x 109/L
* Adequate hepatic function: ALT and AST ≤ 2.5 x ULN, bilirubin ≤ 1.5 x ULN (exception if Gilbert's syndrome ≤ 2.5 x ULN)
* Adequate renal function: calculated creatinine clearance ≥ 50 mL/min, according to the formula of Cockcroft-Gault
* Patient is able to swallow the trial drugs and comply with trial requirements
* Patient agrees not to father a child during participation in the trial and during 3 months thereafter
* Patient agrees to participate to the mandatory translational research part of the trial with exception of Pyruvate dehydrogenase sub-study.

Exclusion Criteria:

* Known or suspected Central nervous system CNS metastases or active leptomeningeal disease
* Previous malignancy within 2 years prior to registration, with the exception of localized non-melanoma skin cancer and Ta and Tis bladder cancer
* Prior treatment for prostate cancer with

  * novel endocrine agents (including abiraterone acetate, enzalutamide, TAK-700, TAK-683, TAK-448, VT464, darolutamide, apalutamide),
  * radioisotopes,
  * TKI and other small molecules,
  * immunotherapy,
  * chemotherapy (with the exception of docetaxel chemotherapy in hormone sensitive prostate cancer)
* Treatment with experimental drugs or treatment within a clinical trial within 30 days prior to registration (except the clinical trial SAKK 96/12, PEACE-4 and/or the biobank project SAKK 63/12)
* Clinically significant cardiovascular disease including:

  * Myocardial infarction within 6 months prior to registration,
  * Uncontrolled angina within 3 months prior to registration,
  * Congestive heart failure NYHA class III or IV,
  * QTc interval > 480 ms,
  * History of clinically significant ventricular arrhythmias (e.g. ventricular tachycardia, ventricular fibrillation, torsades de pointes),
  * History of Mobitz II second or third degree heart block without a permanent pacemaker in place,
  * Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg OR diastolic blood pressure > 105 mmHg
* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment (e.g. uncontrolled or acute severe infection, advanced chronic obstructive pulmonary disease, heart failure)
* Known history of HIV, hepatitis B, hepatitis C
* Major surgery within 4 weeks prior to registration
* Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within 3 months prior to registration)
* Treatment with metformin within the last 6 months prior to registration
* Patients on pharmacotherapy for diabetes mellitus
* History of diabetic ketoacidosis, diabetic coma and pre-coma
* Known history of seizures or any conditions that may predispose to seizure. History of loss of consciousness or transient ischemic attack within 12 months prior to registration
* Concurrent anticoagulation with rivaroxaban or warfarin
* Known hypersensitivity to the IMPs or hypersensitivity to any of their components
* Any concomitant drugs contraindicated for use with the IMPs according to the Swissmedic approved product information
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol and follow-up.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Disease control (DC) | at 15 months
  The primary endpoint of the trial is disease control (DC) at 15 months.

SECONDARY OUTCOMES:
Overall response (OR) | at 15 months
  Overall response (OR) according to modified RECIST and PCWG2 recommendations.
Event-free survival (EFS) | at 15 months
  EFS is defined as the time from randomization until progression or death due to any reason.
Adverse events (AEs) | at 15 months
  AEs will be assessed according to NCI CTCAE v4.0.
Overall survival (OS) | at 15 months
  OS will be calculated from randomization until death due any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rothermundt, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (16):
- Switzerland (16):
  - Kantonsspital Aarau, Aarau
  - Universitaetsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona
  - Kantonsspital Graubuenden, Chur
  - Spital Thurgau AG, Frauenfeld
  - Hôpitaux Universitaires de Genève, Geneva
  - CCAC Lausanne, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Hôpital du Valais, Martigny-Ville
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Hôpital du Valais, Sion
  - Bürgerspital Solothurn, Solothurn
  - Kantonsspital Winterthur, Winterthur
  - Stadtspital Triemli, Zurich
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No